CLINICAL TRIAL: NCT02408991
Title: Proteomics and Stem Cell Therapy as a New Vascularization Strategy
Brief Title: Use Art-assist and Neupogen to Treat Chronic Limb Ischemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left University
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-0553
Record Dates: First submitted 2015-03-13; First posted 2015-04-06 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Lower Limb Ischemia
Keywords: Chronic lower limb ischemia; Art-Assist Device; Neupogen
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AA and Neopogen (Experimental): Patient undergoes treatment with Art-assist device and Neupogen
  Interventions: Drug: Neupogen; Device: Art-Assist Device

INTERVENTIONS:
Drug: Neupogen — Neupogen is given as an injection in your skin every three days for a total of 5 doses.
  Other Names: Filgrastim
Device: Art-Assist Device — The programmed pneumatic compression device (PPCD) is to be worn for a minimum of three hours daily while patient is sitting down
  Other Names: The programmed pneumatic compression device (PPCD)

SUMMARY:
The purpose of this study is to measure the concentration of cells and proteins in the patient's blood during administration of Nuopogen (Filgrastim), a medication that is FDA approved for stem cell mobilization, in combination with a programmed pneumatic compression device (PPCD) (Art-Assist Device). The Art-Assist Device is an FDA approved device that promotes blood flow in the patient's legs. A patient will be prescribed this device and this drug to help improve the poor circulation in his/her leg. The use of Nuopogen along with the Art-Assist Device has not been approved by the FDA and is considered experimental.

This study is not designed to find out how well the Art-Assist Device works, nor how well the drug works in mobilizing stem cells. Instead, it is a study of how well cells lining blood vessels in calf respond to increases in shear stress, and how well the increase in the population of certain cells in the blood stream effect how the new blood vessels will form. It is important for clinical reasons, and for the purposes of this study, that the patient uses the Art-Assist Device as prescribed on a daily basis as discussed with the patient's doctor

DETAILED DESCRIPTION:
This protocol is the next clinical step in our biochemical assessment of a cell therapy approach to treat Chronic Limb Threatening Ischemia (CLI). Briefly, the capability to enlarge collateral arteries ("arteriogenesis"), and to stimulate growth of new capillaries, arterioles and venules at the tissue level ("angiogenesis") is innate. Investigators attribute the failure for this to occur in CLI to the ischemic environment. In our first protocol investigators used an external programmed pneumatic compression device (Art-Assist Device) to improve hemodynamics in the limb and most importantly to provide the "on-switch" to activate the endothelium so arteriogenesis can begin. This new protocol provides the second step in improving this environment; improving the cellular deficit and protein signaling. Investigators are seeking the proteomic, biochemical, and cytometry data needed to refine the approach so a clinical trial can be performed. This project will use FDA approved and CMS reimbursed products.

Rationale

Neovascularization in CLI fails for hemodynamic ("A") and cellular ("B") reasons:

A) The hemodynamic failure caused by multi-level arterial occlusive disease leads to:

1. Attenuation of infra-geniculate endothelial shear stress: Without this stimulus, the endothelial cells lining small collateral arteries are not induced to attract and capture circulating monocytes and progenitor cells that would orchestrate arteriogenesis.
2. Impaired inflow of oxygenated nutritive blood flow into the ischemic tissue
3. Impaired clearance of waste products of metabolism from the ischemic tissue
4. Impaired dissemination of protein signals from the ischemic tissue that would recruit pro-angiogenic reparative cells.
5. Impaired arrival of these pro-angiogenic cells to the ischemic tissue. B) Deficiency in the circulating progenitor cell population: These cells participate in angiogenesis and arteriogenesis. They are deficient in number and in function in CLI patients.

C) Impaired immunity. Even when blood flow is improved there is a population of patients that still succumb to infection. Part of this relates to poor wound management, the other is impaired immunity.

Our cell therapy approach is designed to address each of these. Specifically:

A) The hemodynamic failure caused by multi-level arterial occlusive disease will be corrected by wearing the ACI device that

1. Restores the endothelial shear stress needed to activate vascular endothelium so as to start the Arteriogenesis process.
2. Increases delivery of oxygenated nutritive blood flow into the ischemic tissue
3. Clears waste products of metabolism from the ischemic tissue
4. Increases dissemination of protein signals from the ischemic tissue that would recruit pro-angiogenic reparative cells.
5. Enhances delivery of these pro-angiogenic cells back to the ischemic tissue.

B) The deficiency in the circulating progenitor cell population will be corrected:

G-CSF (Nuopogen, Amgen Inc.) is FDA approved for progenitor/stem cell mobilization. It has been used clinically as stand-alone neovascularization therapy. Investigators will use it in this protocol to correct the deficiency in this vital cell population in CLI patients, enhancing arteriogenesis and angiogenesis. Investigators will measure its biochemical impact.

C) The Impaired immunity will be addressed G-CSF (Nuopogen, Amgen Inc.) is FDA approved for correcting the immunological deficit following cytotoxic chemotherapy. CLI occurs in elderly, often diabetic, patients with impaired immunity. Amputations result when infections arise in the forefoot and reach the mid-foot.

Our hypothesis: is that the combined use of a PPCD and G-CSF will promote arteriogenesis. Investigators have limited but strong clinical evidence that this combined approach dramatically improves blood flow. The recently completed IRB project (IRB#12-1198) focused on the biochemistry of the PPCD. The present submission addresses the biochemical impact of the PPCD and G-CSF together.

B.OBJECTIVES:

Specific Aim 1: is to measure the influence of progenitor cell mobilization on the PPCD proteomic profile investigators derived during our recently completed protocol (IRB # 12-1198). Ten CLI patients will be enrolled. All will wear the PPCD as before. All will receive 10 mcg/kg of Filgrastim (Nuopogen, Amgen Inc.) for a total of 5 doses. The FDA approved indication is stem cell mobilization. The dosimetry is less aggressive than the product label as the dosimetry is being spread out to once every 72 hours rather than once a day. The FDA has granted the PI an IND waiver for this dosing interval. As with our first protocol, cytometry will yield the distribution of progenitor CD34+ and VEGFR2+ cells and monocytes (CD14+). The distribution of mature circulating endothelial cells (CD31+) cells will be measured as a reference point. As with our first protocol investigators will do a proteomic survey measuring levels of cytokines associated with arteriogenesis, as well as serum nitrite (reflection of nitric oxide synthase activity).

Specific Aim 2: investigators will examine the association between these biochemical data, hemodynamic testing, and clinical course (alleviation or progression of forefoot ischemic rest pain and ischemic forefoot wounds) over a 6 month interval.

Study Design: Ten CLI patients with ischemic forefoot rest pain, non-healing forefoot ulceration, or dry forefoot gangrene will be recruited. They will have already undergone standard of care evaluation, including hemodynamic testing and duplex ultrasound delineation of the arterial anatomy in the Non-invasive Vascular Laboratory. Those with tibial artery occlusive disease, with normal or corrected proximal aorto-ilio-femoral arterial anatomy, will be given the option of enrollment in lieu of surgery or catheter revascularization. PPCD use will continue until the presenting symptoms resolve or traditional revascularization becomes necessary to achieve limb salvage. The only three amendments to our first IRB submission (IRB#12-1198) are:

1. All will receive 10 mcg/kg of Filgrastim (Nuopogen, Amgen Inc.) for a total of 5 doses.
2. The 30 day CRC visit will be replaced with a 14 day visit.
3. Cytometry will also be performed on the 14 day visit. As in our first IRB submission, each patient serves as his/her own control. Two "pairs" of blood specimens will be analyzed per patient. A "pair" includes phlebotomy prior to and immediately after two hours of PPCD. The first pair is obtained on enrollment in the CRC. The second pair will be done 2 weeks later 18-24 hours after the last dose of G-CSF. The patient will return for standard of care clinical evaluation, with repeat hemodynamic testing 6 months after that 14 day CRC evaluation.

Baseline visit (Vascular Surgery Clinic):

1. Patients will undergo standard of care history and physical (H&P) examination.
2. Other standard of care tests will include: duplex ultrasound (DUS), Ankle and Toe Pressures.
3. Upon verification that the patient is eligible (based on the inclusion/exclusion criteria), an ICF (Informed consent form), will be explained to the patient to better explain and the study and ask for authorization to participate.

Day1 (at the CRC; Clinical Research Center, University of Chicago): The following procedures will be done in this order:

1. Initial blood draws (20 ml)
2. Each patient will be given Nuopogen shot (10 mcg/kg) subcutaneously.
3. Patients then will wear the PPCD in seated position for (2-hour session).
4. After the 2-hour use of the PPCD, another blood draw will be done (20 ml).
5. Patient will be given ample time to fill out the quality of life questionnaires and the study coordinator will be available at this time to assist the patient.
6. Blood samples will be sent to the Dr. T.C. HE, PhD Lab for analysis.

Days 4, 7, 10, and 13 (at Home or in clinic): The following procedures will be done:

1. Nurse or P.I. will administer Nuopogen shot (10 mcg/kg) subcutaneously, every 3rd day, for a total of 5 Nuopogen shots.
2. Patient will continue use of the PPCD every day, at least 3 hours a day, till symptoms are resolved.

Day14 (at the CRC; Clinical Research Center, University of Chicago): The following procedures will be done in this order:

1. Initial blood drawing (20 ml), 18-24 hours after the 5th shot of Nuopogen. Blood samples will be sent to Dr. T.C. He, PhD Lab for biochemical analysis.
2. Patients will then wear PPCD for 2 hours in seated position.
3. Just prior to the end of the 2-hour use of the PPCD, another blood draw will be done (20 ml).
4. QOL will be filled by the patient.
5. Patient will return the empty vials of Nuopogen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 40 and 85.
2. Chronic limb ischemia Fontaine Class III (ischemic forefoot rest pain) and Class IV (non-healing ischemic ulcers, gangrene) with confirmatory non-invasive vascular testing.

Exclusion Criteria:

1. Acute limb ischemia requiring emergency treatment.
2. Non-salvageable foot (e.g. extensive gangrene, advanced infection, rigor mortis, knee/hip flexion contracture, post-stroke paralysis, and hemiparesis).
3. Untreated hypercoagulability disorder, sickle cell anemia, myeloproliferative disorder.
4. Dialysis, and sustained elevated Creatinine > 4 mg/dl.
5. Severe dementia; bed-ridden; non-compliance; unlikely to follow-up; unreliable.
6. Intolerance of PPCD compression
7. Morbid obesity (Body Mass Index > 34)
8. Severe venous insufficiency causing venous stasis ulceration and dermatitis.
9. Uncorrected significant aorto-iliac, common femoral, and profunda femoral arterial disease
10. Ulceration precluding PPCD placement.
11. Active cancer.
12. Allergy to Nuopogen.
13. Uncorrected symptomatic coronary artery disease
14. History of lymphoma or leukemia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measuring the pharmacologic increase in of CD31+ (mature endothelial cell) | 4 months
  Using the FACSaria sorter. Following clot formation (30 min) each tube will be centrifuged for 15 min at 1000g and the separated serum will be stored at -20° C. Protein will be measured using Enzyme-linked immunosorbent assays (ELISA).

SECONDARY OUTCOMES:
Measureing the pharmacologic increase in CD34+(progenitor cell), | 4 months
  Using the FACSaria sorter. Following clot formation (30 min) each tube will be centrifuged for 15 min at 1000g and the separated serum will be stored at -20° C . Protein will be measured using Enzyme-linked immunosorbent assays (ELISA).
Measureing the pharmacologic increase in VEGFR2+ (endothelial progenitor cell) | 4 months
  Using the FACSaria sorter. Following clot formation (30 min) each tube will be centrifuged for 15 min at 1000g and the separated serum will be stored at -20° C . Protein will be measured using Enzyme-linked immunosorbent assays (ELISA).
Pharmacologix measurement of nitrite | 4 months
  Nitrite will be measured with a quantitative fluorometric assay based on the reaction of nitrite with 2,3- diaminonaphthalene under acidic conditions to form the highly fluorescent 1-(H)-naphthotriazole: 80 l of freshly prepared DAN reagent (25 M in 0.62 M HCl) is added to each 0.8 ml medium sample and mixed immediately. After 10-min incubation at 20°C, the reaction is terminated with 40 l 2.8N NaOH. Formation of 1-(H)-naphthotriazole is measured with a spectrofluorophotometer (model RF-5000; Shimadzu, Kyoto, Japan) with excitation at 380 nm and emission at 405 nm. Nitrite concentrations are determined relative to a standard curve.

CONTACTS AND LOCATIONS:
Overall Officials: Darwin Eton, MD, Principal Investigator — Univ of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bussolino F, Ziche M, Wang JM, Alessi D, Morbidelli L, Cremona O, Bosia A, Marchisio PC, Mantovani A. In vitro and in vivo activation of endothelial cells by colony-stimulating factors. J Clin Invest. 1991 Mar;87(3):986-95. doi: 10.1172/JCI115107. PMID 1705569
- [Background] Bussolino F, Wang JM, Defilippi P, Turrini F, Sanavio F, Edgell CJ, Aglietta M, Arese P, Mantovani A. Granulocyte- and granulocyte-macrophage-colony stimulating factors induce human endothelial cells to migrate and proliferate. Nature. 1989 Feb 2;337(6206):471-3. doi: 10.1038/337471a0. PMID 2464767
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Semerad CL, Christopher MJ, Liu F, Short B, Simmons PJ, Winkler I, Levesque JP, Chappel J, Ross FP, Link DC. G-CSF potently inhibits osteoblast activity and CXCL12 mRNA expression in the bone marrow. Blood. 2005 Nov 1;106(9):3020-7. doi: 10.1182/blood-2004-01-0272. Epub 2005 Jul 21. PMID 16037394
- [Background] Leone AM, Rutella S, Bonanno G, Contemi AM, de Ritis DG, Giannico MB, Rebuzzi AG, Leone G, Crea F. Endogenous G-CSF and CD34+ cell mobilization after acute myocardial infarction. Int J Cardiol. 2006 Aug 10;111(2):202-8. doi: 10.1016/j.ijcard.2005.06.043. Epub 2005 Jul 26. PMID 16051386
- [Background] Takai H, Miyoshi A, Yamazaki M, Adachi K, Katagiri K, Arakawa H, Katsuyama K, Ito T, Fujii E, Hayashi S, Kato A, Suzuki M. Granulocyte colony-stimulating factor has no adverse effects on atherosclerotic lesions in high cholesterol-fed miniature Swine. J Vet Med Sci. 2008 Sep;70(9):943-50. doi: 10.1292/jvms.70.943. PMID 18840969
- [Background] Cavallaro AM, Lilleby K, Majolino I, Storb R, Appelbaum FR, Rowley SD, Bensinger WI. Three to six year follow-up of normal donors who received recombinant human granulocyte colony-stimulating factor. Bone Marrow Transplant. 2000 Jan;25(1):85-9. doi: 10.1038/sj.bmt.1702072. PMID 10654020